CLINICAL TRIAL: NCT04674215
Title: The Effect of Preoperative Turning in Bed and Mobilization Training on the Postoperative First Mobility of Patients Who Will Have Lumbar Disc Surgery
Brief Title: The Effect of Preoperative Turning in Bed and Mobilization Training on the Postoperative First Mobility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi Gulhane Tip Fakultesi (Other)
Responsible Party: Principal Investigator, Hatice Cinar, Doctoral student/Nurse/Principal Investigator, Saglik Bilimleri Universitesi Gulhane Tip Fakultesi
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: YL-20
Record Dates: First submitted 2020-10-06; First posted 2020-12-19 (Actual); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: Postoperative Mobility
Keywords: Postoperative; Nursing; Lumbar Disk Surgery; Role Playing
MeSH Terms: interventions — Beds; Educational Status

STUDY DESIGN:
Intervention Model Description: While the patients receiving control treatment received routine clinical care, the patients in the intervention group received in- bed rotation and mobilization training with planned training with planned training one day before the operation.
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): Data about sociodemographic and clinical characteristics of the patients in all groups were collected. Their mobility status and general anxiety levels were evaluated.
  The patients in the intervention group were given a planned "in-bed turning and mobilization training" in the patient's room by the researcher one day before the surgery. This training included explaining the importance of postoperative mobility, demonstrating the correct in-bed turning and mobilization steps through pictures with the "Illustrated In-Bed Turning and Mobilization Training Material", answering questions (if any), and finally, simulating postoperative in-bed turning and the first mobilization using the role-playing technique in collaboration with the patient.
  Interventions: Behavioral: Turning in Bed; Behavioral: Mobilization; Other: information
- control group (Other): Data about sociodemographic and clinical characteristics of the patients in all groups were collected. Their mobility status and general anxiety levels were evaluated.
  Patients in the control group received routine clinical care. This care included the provision of verbal information to the patient at different times by the primary physician and/or nurse about postoperative in-bed turning and mobilization and answering questions if any.
  Interventions: Other: information

INTERVENTIONS:
Behavioral: Turning in Bed — Preoperative Turning in Bed Training
  Other Names: EDUCATİON
  Arms: intervention group
Behavioral: Mobilization — Preoperative Mobilization Training
  Other Names: EDUCATİON
  Arms: intervention group
Other: information — Routine Clinical Care

SUMMARY:
The purpose of this study is to examine the effect on the first mobility of inside bed rotation and mobilization training to patients who will be lumbar disc surgery.

DETAILED DESCRIPTION:
The purpose of this study is to examine the effect on the first mobility of inside bed rotation and mobilization training to patients who will be lumbar disc surgery. This study Is a randomized controlled clinical trial. The sample of this study consisted of 40 operated with the diagnosis lumbar disc herniation patients that 19 of which were intervention and 21 of which were control patients between January- November 2019. The patients were taken to the table randomization method in the study. While the patients receiving control treatment received routine clinical care, the patients in the intervention group received in- bed rotation and mobilization training with planned training with planned training one day before the operation.

ELIGIBILITY:
Inclusion Criteria:

* Being over the age of 18,
* Being literate in Turkish,
* Being in the ASA(American Society of Anesthesiologists) 1,2 and 3 classification,
* Having surgery for the first time due to lumber disc herniation and volunteering to participate in the research.

Exclusion Criteria:

* Having a mental or physical disability to prevent in-bed rotation and mobilization training to be given before surgery,
* to get a score above 16 from the Observer Mobility Scale before surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-01-02 (Actual); Primary Completion 2019-05-23 (Actual); Study Completion 2019-11-29 (Actual)

PRIMARY OUTCOMES:
Competence during the first postoperative in-bed turning | Operation day (8 hours after surgery)
  The patient's first postoperative in-bed turning, the intensive care nurse scored the patient's dependence-independence status/degree with the in-bed turning section of the Observer Mobility Scale. The Observer Mobility Scale: During the same four activities following the surgery, the patient's dependence-independence status on the nurse is scored between "1- performing the activity independently" and "5-inability to perform the activity despite help". The score that can be obtained from each item varies between 1 and 5, and the total scale score ranges from 4 to 20. Increased scores indicate inadequate movement skills.
Pain during the first postoperative in-bed turning | Operation day (8 hours after surgery)
  The patient scored the degree of the pain during in-bed turning with the related section of the Patient Mobility Scale. The Patient Mobility Scale: The level of pain and difficulty experienced during four activities performed after surgery is evaluated using a 15-cm-wide visual analog. The score that can be obtained from each item varies between 0-15, and the total scale score ranges from 0 to 120. Increased scores indicate an increased level of pain related to the activity.
Strain during the first postoperative in-bed turning | Operation day (8 hours after surgery)
  The patient scored the degree of the strain during in-bed turning with the related section of the Patient Mobility Scale. The Patient Mobility Scale: The level of pain and difficulty experienced during four activities performed after surgery is evaluated using a 15-cm-wide visual analog. The score that can be obtained from each item varies between 0-15, and the total scale score ranges from 0 to 120. Increased scores indicate an increased level of difficulty related to the activity.
Competence during the first postoperative mobilization | On the first postoperative day
  Following the mobilization, the intensive care nurse evaluated the patient's dependence-independence status/degree during the mobilization steps with the Observer Mobility Scale. The Observer Mobility Scale: During the same four activities following the surgery, the patient's dependence-independence status on the nurse is scored between "1- performing the activity independently" and "5-inability to perform the activity despite help". The score that can be obtained from each item varies between 1 and 5, and the total scale score ranges from 4 to 20. Increased scores indicate inadequate movement skills.
Pain during the first postoperative mobilization | On the first postoperative day
  Following the mobilization, the patient evaluated the degree of pain during mobilization with the Patient Mobility Scale. The Patient Mobility Scale: The level of pain and difficulty experienced during four activities performed after surgery is evaluated using a 15-cm-wide visual analog. The score that can be obtained from each item varies between 0-15, and the total scale score ranges from 0 to 120. Increased scores indicate an increased level of pain related to the activity.
Strain during the first postoperative mobilization | On the first postoperative day
  Following the mobilization, the patient evaluated the degree of the strain during mobilization with the Patient Mobility Scale. The Patient Mobility Scale: The level of pain and difficulty experienced during four activities performed after surgery is evaluated using a 15-cm-wide visual analog. The score that can be obtained from each item varies between 0-15, and the total scale score ranges from 0 to 120. Increased scores indicate an increased level of pain related to the activity.

SECONDARY OUTCOMES:
The willingness of the patients for mobilization | On the first postoperative day
  Their willingness for mobilization was evaluated by the intensive care nurse just before the first mobilization by asking the patients and using the Numeric Rating Scale. The scores on the scale range between "0 - I'm not ready for mobilization" and "10 - I feel ready for mobilization" regarding the pre-mobilization willingness.
Anxiety levels of the patients | On the first postoperative day
  Mobilization-related anxiety levels of the patients were evaluated with the Spielberger State Anxiety Inventory filled out by the patient just before and after the first mobilization. The state anxiety scale consists of 20 items. It evaluates the feelings or behaviors experienced by the individual at a certain time or under certain conditions. The trait anxiety scale, on the other hand, requires the individual to describe how they generally feel. It consists of 20 items. The score that can be obtained from the scale ranges between 20 and 80. A high score indicates a high level of anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Hatice Akkaya, Study Director — Saglik Bilimleri Universitesi Gulhane Tip Fakultesi; Hatice Ayhan, Principal Investigator — Saglik Bilimleri Universitesi Gulhane Tip Fakultesi
Locations (1):
- Gulhane Training and Research Hospital, University of Health Sciences, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Should Patients Walk From the Postanesthesia Care Unit to the General Ward After a Lumbar Discectomy? A Randomized Study — https://pubmed.ncbi.nlm.nih.gov/25261141/
- See also: Establishing clinically meaningful severity levels for the Tampa Scale for Kinesiophobia (TSK-13) — https://pubmed.ncbi.nlm.nih.gov/26516705/